CLINICAL TRIAL: NCT04617925
Title: A Phase 2 Study of Belantamab Mafodotin in Patients With Relapsed or Refractory AL Amyloidosis
Brief Title: A Study of Belantamab Mafodotin in Patients With Relapsed or Refractory AL Amyloidosis
Acronym: EMN27
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting European Myeloma Network (Network)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: European Myeloma Network B.V. (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMN27
Record Dates: First submitted 2020-10-20; First posted 2020-11-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: AL Amyloidosis
Keywords: Belantamab mafodotin
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — belantamab mafodotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- belantamab mafodotin (Experimental): Belantamab mafodotin will be administered as an IV infusion at a dose of 2.5 mg/kg every six weeks until progression of disease, unacceptable toxicity or subsequent therapy, for a maximum of eight doses (approximately 12 months), according to the response adapted modifications
  Interventions: Drug: Belantamab mafodotin

INTERVENTIONS:
Drug: Belantamab mafodotin — Belantamab mafodotin will be administered as a monotherapy intravenously at a 2.5 mg/kg calculated dose

SUMMARY:
This is an open-label, multicenter, Phase 2 study in subjects with previously treated patients with light chain (AL) amyloidosis in need for therapy.

Approximately 35 subjects will receive therapy with belantamab mafodotin. Subject participation will include a Screening Phase, a Treatment Phase, a Post-Treatment Observation Phase, and a Long-term Follow-up Phase.

A safety run-in will be conducted in 6 subjects treated with belantamab mafodotin for at least 1 cycle.

According to the two-stage statistical design of the study, an interim analysis of efficacy will occur. If after 15 patients have been enrolled at least 3 complete or very good partial responses have been recorded, the accrual will continue until all planned patients have been enrolled

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AL amyloidosis, confirmed by histology and typed with immunohistochemistry, immunoelectron microscopy or mass spectrometry or if not available, for patients with biopsy confirmed amyloidosis and cardiac involvement alone, if they also have a negative PYP- or DPD-Tc99m bone scan.
2. Previous systemic therapy for AL amyloidosis
3. Patients must be ≥ 18 years of age.
4. ECOG performance status 0, 1 or 2.
5. Mayo stage 1 or Mayo stage 2 or Mayo stage 3A1-3 defined as both cTnT < 0.035 ng/mL (or in place of cTnT the cTnI < 0.10 ng/mL or high sensitivity Troponin T < 54 ng/L) AND simultaneous NT-proBNP ≤ 332 ng/L, OR EITHER above threshold, or BOTH above threshold but with NTproBNP < 8500 ng/L (stage 3A disease)
6. Supine systolic blood pressure ≥ 90 mmHg
7. Measurable disease defined by at least one of the following:

   1. serum free light chain (FLC) ≥2.0 mg/dL (20 mg/L) with an abnormal kappa:lambda ratio or the difference between involved and uninvolved free light chains (dFLC) ≥2mg/dL (20 mg/L).
   2. presence of a monoclonal spike that is ≥0.5 gr/dl.
8. Symptomatic organ involvement (heart, kidney, liver/GI tract, peripheral nervous system).
9. Patient must have adequate organ function, defined as follows:

   System Laboratory Values

   Hematologic:

   Absolute neutrophil count (ANC) ≥1.5 X 109/L Hemoglobin ≥8.0 g/dL Platelets ≥75 X 109/L

   Hepatic:

   Total bilirubin ≤1.5X ULN (Isolated bilirubin ≥1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) ALT ≤2.5 X ULN Renal: eGFR ≥30 mL/min/ 1.73 m2 Cardiac:LVEF (Echo) Clinically asymptomatic patients with ECHO confirmed LVEF ≥25%
10. Written informed consent in accordance with local and institutional guidelines.
11. Female patients: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies

    A female patient is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:
    * Is not a woman of childbearing potential (WOCBP) OR
    * Is a WOCBP and using a contraceptive method that is highly effective (failure rate of <1% per year), preferably with low user dependency (as described in Appendix 3), during the intervention period and for at least four months after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

    A WOCBP must have a negative highly-sensitive serum pregnancy test (as required by local regulations) within 72 hours before the first dose of study intervention.

    The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with a nearly undetected pregnancy.

    Nonchildbearing potential is defined as follows (by other than medical reasons):
    * ≥45 years of age and has not had menses for >1 year,
    * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation,
    * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.
12. Male Patients : contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

    Male Patients are eligible to participate if they agree to the following during the intervention period and for 6 months after the last dose of study treatment to allow for clearance of any altered sperm:

    • Refrain from donating sperm

    PLUS either:

    • Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent.

    OR

    • Must agree to use contraception/barrier as detailed below: Agree to use a male condom, even if they have undergone a successful vasectomy, and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year as when having sexual intercourse with a WOCBP who is not currently pregnant.
13. All prior treatment-related toxicities (defined by National Cancer Institute- Common Toxicity Criteria for AEs (NCI-CTCAE), version 5, corneal toxicities are defined according to the Keratopathy Visual Activity [KVA] scale) must be ≤ Grade 1 at the time of enrolment except for alopecia.
14. Patients must be able to understand the study procedures and agree to participate in the study by providing written informed consent

Exclusion Criteria:

1. Presence of non-AL amyloidosis.
2. Presence of lytic bone lesions or active myeloma with hypercalcemia, cast nephropathy, anemia due to marrow infiltration or extramedullary disease.
3. Previously untreated disease: patients must have had at least 2 cycles of therapy directed against the plasma cell clone; however, patients that have received high dose therapy with melphalan as their only therapy are eligible for the study.
4. Previous exposure to anti-BMCA agents
5. Cardiac stage IIIB disease: both cTnT > 0.035 ng/mL (or in place of cTnT the cTnI > 0.10 ng/mL or high sensitivity Troponin T > 54 ng/L) AND simultaneous NT-proBNP >8500 ng/L.
6. Known repetitive ventricular arrhythmias on 24h Holter Electrocardiogram (ECG) in spite of anti-arrhythmic treatment. Patients must not have evidence of cardiovascular risk including any of the following:

   * Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant ECG abnormalities such as 2nd degree (Mobitz Type II) or 3rd degree atrioventricular (AV) block.
   * History of myocardial infarction, acute coronary syndromes (including unstable or uncontrolled angina), coronary angioplasty, or stenting or bypass grafting within three (3) months of Screening.
   * Class III or IV heart failure as defined by the New York Heart Association functional classification system [NYHA, 1994]
   * Severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless patient has a pacemaker.
   * Uncontrolled hypertension or hypotension (i.e., supine SBPN < 90 mmHg despite supportive therapy with midodrine)
7. Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 14 days prior to Cycle 1 Day 1.
8. Pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to Cycle 1 Day 1.
9. Current corneal epithelial disease except mild changes in corneal epithelium.
10. Current unstable liver or biliary disease defined by the presence of large volume ascites requiring paracentesis, encephalopathy, coagulopathy, hypoalbuminemia (except due to AL related nephrotic syndrome), esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement due to AL amyloidosis is acceptable if otherwise meets entry criteria.
11. Presence of active renal condition (infection, requirement for dialysis or any other condition that could affect the patient's safety) unrelated to AL amyloidosis. Patients with isolated proteinuria resulting from AL are eligible, provided they fulfil other inclusion criteria
12. Patients must not use contact lenses while participating in this study.
13. Patients must not be simultaneously enrolled in any interventional clinical trial.
14. Use of an investigational drug or approved systemic anti-myeloma therapy (including systemic steroids) within 14 days or five half-lives, whichever is shorter, preceding the first dose of study drug.
15. Plasmapheresis within 7 days prior to first dose of study treatment.
16. Treatment with a monoclonal antibody within 30 days of receiving the first dose of study drugs.
17. Major surgery ≤ 4 weeks prior to initiating study treatment.
18. Any evidence of active mucosal or internal bleeding.
19. Known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to blmf or drugs chemically related to blmf, or any of the components of the study treatment.
20. Active infection requiring treatment.
21. Known HIV infection (defined by positive testing for human immunodeficiency virus (HIV) antibodies).
22. Positive test of hepatitis B surface antigen, or hepatitis B core antibody at screening or within 3 months prior to first dose of study treatment.
23. Positive hepatitis C antibody test result or positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment.

    Note: Patients with positive hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative hepatitis C RNA test is obtained.

    Note: Hepatitis RNA testing is optional and patients with negative hepatitis C antibody test are not required to also undergo hepatitis C RNA testing.
24. Invasive malignancies other than disease under study, unless the second malignancy has been medically stable for at least 2 years and, in the opinion of the principal investigators, will not affect the evaluation of the effects of clinical trial treatments on the currently targeted malignancy. Patients with curatively treated non-melanoma skin cancer may be enrolled without a 2-year restriction.
25. Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including lab abnormalities) that could interfere with the patient's safety, obtaining informed consent or compliance to the study procedures.
26. Patients must not be pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
response rate | at 6 months (cycle 4)
  Complete Response (CR)/ Very Good Partial Response (VGPR)/ <50 mg/L difference between involved minus uninvolved serum free lights chains (low-dFLC) according to the consensus recommendations for AL amyloidosis treatment response criteria

SECONDARY OUTCOMES:
Adverse events | up to 70 days after last dose
  Rates of grade 3 or higher AEs related to blmf therapy
Treatment discontinuation | up to 1 year
  Rates of treatment discontinuation due to toxicity related to blmf
Dose reduction | up to 1 year
  Dose reduction due to toxicity of blmf therapy
Hematologic AEs | up to 70 days after last dose
  rates of any hematologic adverse events
Non-hematologic AEs | up to 70 days after last dose
  rates of any non-hematologic adverse events
Ocular toxicity | up to 1 year
  rates of adverse events of special interest
Overall hematologic response rates | 3 months, 6 months
  Complete Response (CR)/ Very Good Partial Response (VGPR)/ <50 mg/L difference between involved minus uninvolved serum free lights chains (low-dFLC)/ Partial Response (PR)
Organ response rates | 3,6,12,18, and 24 months
  Organ response rates per individual organ (heart, kidney, liver) according to International Amyloidosis Consensus Criteria
Duration of response | approximately up to 9 years
  Duration of response is defined as the time between first documentation of response (achievement of at least a PR or lowdFLC response) and PD
Determine time to progression | approximately up to 9 years
  From the date of registration to the date of first disease progression, major organ deterioration or death, whichever occurs first
Overall survival | approximately up to 9 years
  Overall Survival, measured from the date of from randomization to the date the subject's death

CONTACTS AND LOCATIONS:
Locations (6):
- Centre hospitalier Universitaire de Limoges -, Limoges, France
- University Hospital Heidelberg, Heidelberg, Germany
- General Hospital of Athens "Alexandra", Athens, Greece
- Fondazione I.R.C.C.S Policlinico "San Matteo", Pavia, Italy
- UMC Utrecht, Utrecht, Netherlands
- Royal Free Hospital - London,, London, United Kingdom